CLINICAL TRIAL: NCT06490562
Title: A Prospective Multicenter Randomized Controlled Clinical Trial Protocol for the Efficacy and Safety of Low-dose Cyclophosphamide or CNI in the Prevention of Acute Graft-versus-host Disease After gDLI
Brief Title: Low-dose Cyclophosphamide or CNI in the Prevention of Acute Graft-versus-host Disease After gDLI
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IIT2024034
Record Dates: First submitted 2024-06-19; First posted 2024-07-08 (Actual); Last update posted 2024-07-08 (Actual); Status verified 2024-05

CONDITIONS: Acute Graft-versus-host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PDCy group (Other): Low dose Cy 30 mg/kg/d was administered on the 3rd and 4th day after gDLI to prevent GVHD
  Interventions: Drug: PDCy
- Non Cy group (Other): Oral administration of low-dose CNI (CSA 25mg Q12H or FK506 0.25mg Q12H combined with azole fungal drugs) for 2 weeks to prevent GVHD at 0 days after gDLI
  Interventions: Drug: Non Cy

INTERVENTIONS:
Drug: PDCy — Low dose Cy 30 mg/kg/d was administered on the 3rd and 4th day after gDLI to prevent GVHD
  Arms: PDCy group
Drug: Non Cy — Oral administration of low-dose CNI (CSA 25mg Q12H or FK506 0.25mg Q12H combined with azole fungal drugs) for 2 weeks to prevent GVHD at 0 days after gDLI
  Arms: Non Cy group

SUMMARY:
Assess the cumulative incidence of severe (III-IV) aGVHD after low-dose cyclophosphamide or CNI is used to after gDLI. Evaluate the overall survival rate (OS), non recurrent mortality rate (NRM), and recurrence rate (CIR) of two groups of patients; The complete response rate (CR) and partial response rate (PR) of patients with morphological/extramedullary recurrence, as well as the complete response rate and MRD response rate of patients with molecular recurrence. The incidence of adverse events such as infection, hemorrhagic cystitis, and cardiac events in two groups.

DETAILED DESCRIPTION:
Assess the cumulative incidence of severe (III-IV) aGVHD after low-dose cyclophosphamide or CNI is used to after gDLI. Evaluate the overall survival rate (OS), non recurrent mortality rate (NRM), and recurrence rate (CIR) of two groups of patients; The complete response rate (CR) and partial response rate (PR) of patients with morphological/extramedullary recurrence, as well as the complete response rate and MRD response rate of patients with molecular recurrence. The incidence of adverse events such as infection, hemorrhagic cystitis, and cardiac events in two groups.

Efficacy Evaluation: Follow up observation of the difference in efficacy and safety between two groups in preventing severe (III-IV) aGVHD.

Primary Exploratory Endpoint: Assess the cumulative incidence of severe (III-IV) aGVHD after low-dose cyclophosphamide or CNI is used after gDLI.

Secondary Exploratory Endpoints:

1. 1-year overall survival rate (OS);
2. 1-year recurrence rate (CIR);
3. 1-year non recurrent mortality rate (NRM);
4. The complete response rate (CR) and partial response rate (PR) of patients with morphological/extramedullary recurrence, as well as the complete response rate and MRD response rate of patients with molecular recurrent minimal residual disease (MRD);
5. The incidence of adverse events such as infection, hemorrhagic cystitis, and cardiac events in two groups.

ELIGIBILITY:
Inclusion Criteria:

* Subjects eligible for inclusion in this study must meet all of the following criteria:

  1. Patients with malignant hematological diseases undergo haploid/sibling incomplete matching/unrelated donor transplantation;
  2. Recurrence after transplantation (morphological, extramedullary, or molecular recurrence);
  3. Plan to administer granulocyte colony-stimulating factor mobilization donor lymphocyte infusion (gDLI) for treatment;
  4. No age, gender, or race restrictions;
  5. The physical condition assessment (ECOG-PS) of the Eastern Oncology Collaborative Group is 0-2 points;
  6. The patient or their authorized representative agrees to participate in the clinical trial and signs an informed consent form.

Exclusion Criteria:

* Subjects meeting any of the following criteria are not eligible for inclusion in this study:

  1. Siblings of matched donor transplant;
  2. Patients with other malignant tumors that require treatment;
  3. There are active infections, such as hepatitis B, hepatitis C, tuberculosis, etc;
  4. HIV serological reaction was positive;
  5. Suffering from mental illness or other conditions that cannot comply with research, treatment, and monitoring requirements;
  6. Pregnant patients or patients who are unable to take appropriate contraceptive measures during treatment;
  7. Active heart disease is defined as one or more of the following:

     1. Have a history of uncontrolled or symptomatic angina pectoris;
     2. Myocardial infarction less than 6 months prior to enrollment in the study;
     3. A history of arrhythmia requiring medication treatment or severe clinical symptoms;
     4. Uncontrolled or symptomatic congestive heart failure (>NYHA level 2);
     5. The ejection fraction is below the lower limit of the normal range.
  8. Individuals who are allergic to any medication or component such as Cy, CNI, etc;
  9. The researchers believe that it is not suitable for participants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Assess the cumulative incidence of severe (III-IV) aGVHD after low-dose cyclophosphamide or CNI is used after gDLI. | Until the end of the study
  Assess the cumulative incidence of severe (III-IV) aGVHD after low-dose cyclophosphamide or CNI is used after gDLI.

SECONDARY OUTCOMES:
1-year overall survival rate (OS) | 1 year after the last patient was enrolled
  1-year overall survival rate (OS)
1-year recurrence rate (CIR) | 1 year after the last patient was enrolled
  1-year recurrence rate (CIR)
1-year non recurrent mortality rate (NRM) | 1 year after the last patient was enrolled
  1-year non recurrent mortality rate (NRM)
The complete response rate (CR) and partial response rate (PR) of patients with morphological/extramedullary recurrence, as well as the complete response rate and MRD response rate of patients with molecular recurrent minimal residual disease (MRD) | 1 year after the last patient was enrolled
  The complete response rate (CR) and partial response rate (PR) of patients with morphological/extramedullary recurrence, as well as the complete response rate and MRD response rate of patients with molecular recurrent minimal residual disease (MRD)
The incidence of adverse events such as infection, hemorrhagic cystitis, and cardiac events in two groups. | 1 year after the last patient was enrolled
  The incidence of adverse events such as infection, hemorrhagic cystitis, and cardiac